CLINICAL TRIAL: NCT04062136
Title: Outcomes of Human Umbilical Cord-derived Mesenchymal Stem Cells Transplantation in the Treatment of Bronchopulmonary Dysplasia
Brief Title: Umbilical Cord Mesenchymal Stem Cells Transplantation in the Treatment of Bronchopulmonary Dysplasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VinmecISC1915
Record Dates: First submitted 2019-03-27; First posted 2019-08-20 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary dysplasia; umbilical cord mesenchymal stem cells
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stem cell transplantation (Experimental): 1 million umbilical Cord Mesenchymal Stem Cells per body kg will transplant via the intravenous at baseline, and the second transplantation will be performed 1 week after the first transplantation
  Interventions: Combination Product: stem cell transplantation

INTERVENTIONS:
Combination Product: stem cell transplantation — Transplantation of umbilical cord mesenchymal stem cells

SUMMARY:
To evaluate the safety and efficacy of human umbilical cord mesenchymal stem cells transplantation in patients with bronchopulmonary dysplasia

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and effectiveness of human umbilical cord mesenchymal stem cells in 10 patients with bronchopulmonary dysplasia at Vinmec International Hospital, Hanoi, Vietnam

ELIGIBILITY:
Inclusion Criteria:

* The patient is diagnosis Bronchopulmonary Dysplasia (premature and depends on oxygen until 28 days old
* Gender: either sex
* Year old < 6 months
* Weight ≥ 2 kg
* Agree to participate in the study.

Exclusion Criteria:

* Severe congenital malformation.
* Other severe conditions (active pulmonary bleeding, evidence of active infections).

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events | during 9 months post treatment
  Incidence of the adverse events or serious adverse events after transplantation
The proportion of patients win from oxygen | during 9 months post treatment
  To identify the proportion of patient with Bronchopulmonary Dysplasia win from oxygen after stem cell transplantation.

SECONDARY OUTCOMES:
The lung fibrosis | at 6 months post treatment
  Changes of the lung fibrosis on chest CT at 6 months compared with baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahn SY, Chang YS, Kim SY, Sung DK, Kim ES, Rime SY, Yu WJ, Choi SJ, Oh WI, Park WS. Long-term (postnatal day 70) outcome and safety of intratracheal transplantation of human umbilical cord blood-derived mesenchymal stem cells in neonatal hyperoxic lung injury. Yonsei Med J. 2013 Mar 1;54(2):416-24. doi: 10.3349/ymj.2013.54.2.416. PMID 23364976
- [Result] Chang YS, Ahn SY, Yoo HS, Sung SI, Choi SJ, Oh WI, Park WS. Mesenchymal stem cells for bronchopulmonary dysplasia: phase 1 dose-escalation clinical trial. J Pediatr. 2014 May;164(5):966-972.e6. doi: 10.1016/j.jpeds.2013.12.011. Epub 2014 Feb 6. PMID 24508444
- [Result] Liem NT, Anh TL, Thai TTH, Anh BV. Bone Marrow Mononuclear Cells Transplantation in Treatment of Established Bronchopulmonary Dysplasia: A Case Report. Am J Case Rep. 2017 Oct 12;18:1090-1094. doi: 10.12659/ajcr.905244. PMID 29021519